CLINICAL TRIAL: NCT03958058
Title: Tick-Borne Encephalitis Virus and Lyme Borreliae Causing Coillness, Coinfection, or Just Coincidence. A Prospective Observational Study
Brief Title: Tick-borne Encephalitis and Possible Borrelial Serology
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana School of Medicine, Slovenia (Other)
Responsible Party: Principal Investigator, Daša Stupica, Prinicipal Investigator, University Medical Centre Ljubljana
Other Study IDs: TBE-LB observational
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Tick Borne Encephalitis; Lyme Disease
MeSH Terms: conditions — Encephalitis, Tick-Borne; Lyme Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anti-borrelial antibiotic therapy
  Interventions: Drug: Anti-borrelial antibiotic therapy
- No antibiotics: Patients who received symptomatic therapy (paracetamol, Lekadol®, granisetron, Kytril®, metamizol, Analgin®, parenteral hydration with saline). Patients reported the presence of nonspecific symptoms such as headache, fatigue, arthralgia, myalgia.
  Interventions: Other: No antibiotic.

INTERVENTIONS:
Drug: Anti-borrelial antibiotic therapy — Beside symptomatic therapy, patients received oral doxycycline 100 mg (Doxy®) twice daily or ceftriaxone 2 g (Lendacin®) once daily for 14 days. Antibiotic therapy was left to the discretion of treating physicians. Patients reported the presence of nonspecific symptoms such as headache, fatigue, arthralgia, myalgia.
  Groups: Anti-borrelial antibiotic therapy
Other: No antibiotic. — Patients who received symptomatic therapy (paracetamol, Lekadol®, granisetron, Kytril®, metamizol, Analgin®, parenteral hydration with saline). Patients reported the presence of nonspecific symptoms such as headache, fatigue, arthralgia, myalgia.
  Groups: No antibiotics

SUMMARY:
In Europe, tick-borne encephalitis (TBE) virus causing TBE is transmitted by the bite of Ixodes ricinus tick, which can also transmit Lyme borreliae , the causative agent of Lyme borreliosis (LB). Since TBE and LB are both endemic with high incidence rates in Slovenia, we should be attentive to the possibility of double infections. Double infections with TBE virus and Lyme borreliae were reported to occur rarely even in endemic countries, however reliable data on coinfection rates are rather limited. Microbiological diagnosis of TBE virus infection is quite straightforward, and there is no specific therapy for TBE available so far. This markedly differs from borrelial infection, in which case interpretation of serological test results demands more caution, but there is highly efficient antibiotic treatment available for LB. This may lead to over prescribing of antibiotics to TBE patients with documented borrelial antibodies in serum indicating possible coinfection with Lyme borreliae, but missing clinical or microbiological criteria for proven borrelial coinfection. Approximately 10% of patients who had been treated appropriately for LB and about one third of patients after TBE report nonspecific subjective complaints, such as fatigue, headache, arthralgia, and myalgia, termed post-Lyme and post-encephalitic symptoms, respectively. These may not be differentiated clearly from nonspecific symptoms occurring with a rather substantial incidence also in the general population. A trend of ascribing medically unexplained nonspecific subjective symptoms to LB in subjects with positive borrelial antibodies in serum puzzles the situation further.

The aim of this prospective observational study was to assess the proportion and clinical implication of proven and possible coinfection with Lyme borreliae in patients with TBE, and to evaluate the association between anti-borrelial antibiotic therapy and clinical outcome in the subgroup of patients with possible coinfection.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* admitted between January 2007 and December 2013 at the University Medical Centre Ljubljana, Slovenia
* tick-borne encephalitis defined according to European criteria (febrile illness with symptoms and/or signs of meningitis or meningoencephalitis, cerebrospinal fluid (CSF) pleocytosis (>5 × 106 cells/L), and demonstration of acute TBE virus infection (the presence of specific tick-borne encephalitis virus IgM and IgG antibodies in serum or demonstration of intrathecal production of specific TBE virus IgM and/or IgG antibodies in patients previously vaccinated against tick-borne encephalitis)

Exclusion Criteria:

* Lyme borreliosis in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with tick-borne encephalitis.
Sampling Method: Non-Probability Sample
Enrollment: 690 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with objective manifestations of Lyme borreliosis | up to 12 months follow-up
  At each visit physical examination was performed and clinical signs indicating objective manifestations of Lyme borreliosis, such as erythema migrans, were searched for and documented.
Frequency of nonspecific symptoms such as headache, fatigue, arthralgia, myalgia | up to 12 months follow-up
  At each visit patients were asked to report the presence of nonspecific symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia